CLINICAL TRIAL: NCT01827657
Title: A Phase I, Open-Label, Parallel-Group, Two-Part Study to Evaluate the Pharmacokinetics and Safety of GSK2336805 in Subjects With Hepatic Impairment and Healthy Matched Control Subjects (HAI117380)
Brief Title: Study to Evaluate the Pharmacokinetics and Safety of GSK2336805 in Subjects With Hepatic Impairment and Healthy Matched Control Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117380
Record Dates: First submitted 2013-04-05; First posted 2013-04-09 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis C
Keywords: plasma; tolerability; safety; matched control; GSK2336805; hepatic impairment; pharmacokinetics
MeSH Terms: conditions — Hepatitis C | interventions — GSK2336805

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 Cohort 1 - Mild hepatic impairment (Experimental): Subjects with mild hepatic impairment will be enrolled in Cohort 1 and will receive a single dose of 60 mg GSK2336805
  Interventions: Drug: GSK2336805
- Part 1 Cohort 2 - Moderate hepatic impairment (Experimental): Subjects with moderate hepatic impairment will be enrolled in Cohort 2 and will receive a single dose of 60 mg GSK2336805
  Interventions: Drug: GSK2336805
- Part 1 Cohort 3 - Matched healthy volunteers to Cohort 2 (Experimental): Control subjects will be matched for gender, age (+/- 10 years), body mass index (BMI) (+/- 20%), and smoking status to the subjects in the moderate hepatic impairment arm. These healthy volunteers will receive a single dose of 60 mg GSK2336805
  Interventions: Drug: GSK2336805
- Part 2 Cohort 4 - Severe hepatic impairment (Experimental): Subjects with severe hepatic impairment will be enrolled in Cohort 2 and will receive a single dose of 60 mg GSK2336805. The decision to move forward into Part 2 (severe hepatic impairment) will be based on a review of the preliminary safety and pharmacokinetic data from subjects with moderate hepatic impairment
  Interventions: Drug: GSK2336805
- Part 2 Cohort 5 - Matched healthy volunteers to Cohort 4 (Experimental): Based on emerging data from Part 1, the sponsor may decide to enroll matched controls to the severe hepatic group (i.e. in case of a change in dose or the demographics of the severe hepatic group are not well matched with the moderate control data). The subjects in this optional control cohort will be matched for gender, age (+/- 10 years), BMI (+/- 20%), and smoking status to the subjects in the severe hepatic impairment category
  Interventions: Drug: GSK2336805

INTERVENTIONS:
Drug: GSK2336805 — Two 30 mg GSK2336805 tablets for a 60 mg single dose will be administered in this study

SUMMARY:
This is a single-dose, open-label, two part, parallel group study. This study is being conducted to determine the pharmacokinetics, safety and tolerability of GSK2336805 in subjects with varying degrees of hepatic impairment. Part 1 of the study will enroll subjects with mild and moderate hepatic impairment and healthy control subjects matched to the subjects in the moderate hepatic impairment category. The decision to commence Part 2 will be based on a review of the preliminary safety and pharmacokinetic data from subjects with moderate hepatic impairment. Part 2 will enroll subjects with severe hepatic impairment. Additionally, based on emergent data from Part 1, matched controls to the severe hepatic group may be enrolled (optional). Due to the potential difficulty in identifying eligible subjects with severe hepatic impairment, the study may be stopped prior to full enrollment in Part 2, provided that a minimum of 4 evaluable subjects with severe hepatic impairment have been enrolled. The study will consist of a Screening visit, a single dose Treatment Period and a Follow-up visit. Subjects will be screened for eligibility criteria within 30 days of enrolment. Subjects will be admitted to the clinical unit on Day -1; each subject will receive a single dose of GSK2336805 on Day 1 and will remain in the clinical unit for 5 days (check-out on Day 4). The follow-up visit will be conducted within 7-10 days after Day 1 dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 74 years inclusive, at the time of signing the informed consent.
* Body weight >=45 kilogram (kg) for men and women and body mass index (BMI) within the range 17- 41 kg/meter square (m^2) for hepatically impaired subjects; healthy matched control subjects will be matched to BMI +/- 20% and must also remain in the BMI range of 17- 41 kg/m^2.
* A female subject is eligible to participate if she is of non-childbearing potential (postmenopausal defined as 12 months of spontaneous amenorrhea or pre-menopausal females with a documented tubal ligation or hysterectomy).
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned.
* Ability and willingness to abstain from alcohol-containing beverages/foods from 48 hours prior to entry in the clinical study centre until discharge.
* Supplemental inclusion criteria for Healthy Volunteer subjects only: A male or female is eligible for study participation if he/she is healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and electrocardiogram (ECG), including no cardiac, pulmonary, hepatic, biliary, gastrointestinal, or renal disorders (defined as serum creatinine >1.5 milligram(mg)/decilitre (dL) or a calculated creatinine clearance (CrCl)<50 millilitre (mL)/ minute(min), or cancer within the past 5 years (except localized or in situ cancer of the skin). A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. A single repeat laboratory evaluation is allowed for eligibility determination. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, and bilirubin less than the upper limits of normal. The subject's systolic blood pressure is inside the range of 90-140 millimeter of mercury (mmHg) and diastolic blood pressure is inside the range of 45-90 mmHg and heart rate is inside the range of 50-100 beats per minute (bpm) for female subjects or 45-100 bpm for male subjects.
* Supplemental inclusion criteria for all hepatically impaired subjects: Chronic (>6 months), stable (no acute episodes of illness within the previous 1 month prior to screening due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology. Subjects must also remain stable throughout the Screening period.
* Subjects whose platelets are greater than or equal to 30,000 x 10^9/Liter of blood who have not had any major bleeding episodes within the past 6 months.
* Supplemental inclusion criteria for all hepatically impaired subjects in the mild group: A male or female is eligible for study participation if he/she is considered to have mild hepatic insufficiency (of any etiology) and has been clinically stable for at least 1 month prior to screening. To be classified as having mild hepatic insufficiency, subjects must have: A Child-Pugh score of 5-6 with known medical history of liver disease (with or without a known history of alcohol abuse) and previous confirmation of liver cirrhosis by liver biopsy or other medical imaging technique (including laparoscopy, computed tomography [CT] scan, Magnetic Resonance Imaging [MRI] or ultrasonography) associated with an unambiguous medical history.
* Supplemental inclusion criteria for all hepatically impaired subjects in the moderate group: A male or female is eligible for study participation if he/she is considered to have moderate hepatic insufficiency (of any etiology) and has been clinically stable for at least 1 month prior to screening. To be classified as having moderate hepatic insufficiency, subjects must have: A Child-Pugh score of 7-9 with known medical history of liver disease (with or without a known history of alcohol abuse) and previous confirmation of liver cirrhosis by liver biopsy or other medical imaging technique (including laparoscopy, CT scan, MRI or ultrasonography) associated with an unambiguous medical history.
* Supplemental inclusion criteria for all hepatically impaired subjects in the severe group: A male or female is eligible for study participation if he/she is considered to have severe hepatic insufficiency (of any etiology) and has been clinically stable for at least 1 month prior to screening. To be classified as having severe hepatic insufficiency, subjects must have: A Child-Pugh score of >9 with known medical history of liver disease (with or without a known history of alcohol abuse) and previous confirmation of liver cirrhosis by liver biopsy or other medical imaging technique (including laparoscopy, CT scan, MRI or ultrasonography) associated with an unambiguous medical history

Exclusion Criteria:

* Pregnant females as determined by positive serum or urine Human Chorionic Gonadotropin (hCG) test at screening or prior to dosing.
* Lactating females.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, satsuma, ugli, tangerine, and tangelo, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Use of prescription or non-prescription drugs, vitamins, and herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication. Hepatically impaired subjects requiring prescription or non-prescription drugs may be acceptable provided the medications are not on the Prohibited Medications List of the protocol and in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. In addition, if heparin is used during pharmacokinetic (PK) sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines. For hepatically impaired subjects, a positive drug screen will be allowed if it is due to a prescribed medication, provided that medication is not on the Prohibited Medications List of the protocol.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate <45 and >100 beats per minute (bpm) (males) and <50 and >100 bpm (females); PR Interval <120 and >220 milliseconds (msec); QRS duration <70 and >120 msec; corrected QT interval by Bazett's formula (QTcB) >450 msec or >480 msec in subjects with incomplete Bundle Branch Block; Evidence of previous ischemic, valvular, or congenital heart disease (Does not include ST segment changes associated with repolarization); Any clinically significant conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome); Sinus Pauses >3 seconds; Any significant arrhythmia which, in the opinion of the principal investigator, will interfere with the safety for the individual subject; and Non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats).
* Supplemental exclusion criteria for healthy volunteer subjects only: A positive Hepatitis B surface antigen or positive Hepatitis C antibody result at screening. Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of inflammatory bowel disease should be excluded. Subjects with a history of peptic ulceration or pancreatitis within the preceding 6 months of screening should be excluded. Subjects with any previous gastrointestinal (GI) surgery (except appendectomy or gall bladder removal more than three months prior to study) may be enrolled in this study only if, in the opinion of the Investigator and the Medical Monitor, it is not expected to interfere with the study procedures or to pose an additional safety risk to the subject. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Supplemental exclusion criteria for hepatically impaired subjects only:
* Evidence of recent, acute infection with Hepatitis B and/or Hepatitis C within preceding 6 months. Subjects with chronic Hepatitis B or C (duration >6 months) are eligible for enrolment.
* Subjects with a pre-existing condition (except hepatic impairment) interfering with normal gastrointestinal anatomy or motility that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of inflammatory bowel disease should be excluded. Subjects with a history of peptic ulceration or pancreatitis within the preceding 6 months of screening should be excluded. Subjects with previous gastrointestinal (GI) surgery (except appendectomy or gall bladder removal more than three months prior to study) may be enrolled in this study only if, in the opinion of the Investigator and the Medical Monitor, it is not expected to interfere with the study procedures or to pose an additional safety risk to the subject.
* Subjects receiving lactulose who are medically unable to halt lactulose administration from 8 hour (h) before dosing with study drug to 4h after dosing with study drug.
* Subjects with severe encephalopathy (grade 3 or 4) as judged by the investigator or significant Central Nervous System (CNS) disease (e.g. dementia, or seizures) which the investigator considers will interfere with the informed consent, conduct, completion, or results of this trial or constitutes an unacceptable risk to the subject.
* Subjects with a change in dose regimen of medically required medication within the 2 weeks prior to dosing.
* Subjects with creatinine clearance <=50 mL/min (calculated by the Cockcroft-Gault Formula). If the result calculated by Cockcroft-Gault is between 40 and 50 mL/min, then the site may complete a 24 hour urine collection to more specifically calculate the CrCl. A CrCl value < or = 50mL/min via 24-hour urine collection is also exclusionary.
* History of gastric or esophageal variceal bleeding within the past 6 months and for which varices have not been adequately treated with medication and/or surgical procedures.
* Subjects with electrolyte imbalance whose serum sodium levels are less than or equal to 125 millimol/litre (mmol/L); potassium levels are less than or equal to 2.5 mmol/L; calcium levels less than or equal to 6.1mmol/L).
* Presence of hepatopulmonary or hepatorenal syndrome.
* Primarily cholestatic liver diseases.
* History of liver transplantation.
* Subjects in the severe hepatic impairment group that are expecting a liver transplant during the study participation period.
* Subjects with signs of active bacterial infection (including active spontaneous bacterial peritonitis).
* Subjects with Transjugular Intrahepatic Portosystemic Shunt (TIPS) placement within the past 3 months.
* Subjects with unstable cardiac function or subjects with hypertension whose blood pressure that is not well controlled (based on the investigator's discretion)
* Diabetic subjects whose diabetes that is not controlled (based on the investigator's discretion).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-05-28 (Actual); Primary Completion 2014-03-20 (Actual); Study Completion 2014-03-20 (Actual)

PRIMARY OUTCOMES:
Composite of plasma pharmacokinetic (PK) parameters of GSK2336805 | Day 1: 0.25 hours (h) predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 (Day 2), 36, 48(Day 3), 60 and 72(Day 4) h post-dose
  The following pharmacokinetic parameters will be determined: area under the plasma concentration time curve (AUC)- from time zero to infinity [AUC(0-inf)], from time zero to the last quantifiable time points [AUC(0-t)], and from time zero to 24 hours [AUC(0-24)]; maximum observed plasma concentration (Cmax); time to Cmax (tmax); concentration at 24hour post-dose (C24); absorption lag time (tlag); apparent oral clearance (CL/F), apparent volume of distribution after oral administration (Vz/F), and half-life (t½). These will be compared in subjects with hepatic impairment to healthy volunteers

SECONDARY OUTCOMES:
Safety and tolerability of GSK2336805 as assessed by adverse events (AEs), concurrent medications, clinical laboratory, electrocardiograms (ECGs) and vital sign parameters | Up to 10 days
  Safety and tolerability assessment will include assessment of AEs, concurrent medications, clinical laboratory, ECGs and vital sign
Unbound concentration and unbound fraction of GSK2336805 in plasma | Day 1: 2, 12 and 24 h post dose
  Impact of hepatic impairment on pharmacokinetics of GSK2336805 will be assessed by evaluation of unbound concentration and unbound fraction of GSK2336805 in plasma.
Composite of plasma PK parameters of GSK2336805 in subjects with hepatic impairment compared with PK parameters of non-cirrhotic subjects with chronic Hepatitis C (CHC) | Day 1: 0.25 hours (h) predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 (Day 2), 36, 48 (Day 3), 60 and 72 (Day 4) h post-dose
  The PK parameters: AUC(0-t), AUC(0-inf), Cmax, C24, t½, CL/F, and Vz/F in subjects with hepatic impairment will be compared with PK parameters of non-cirrhotic subjects with CHC in previous studies (HAI114885 and HAI115519)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Knoxville, Tennessee

REFERENCES:
- See also: Results for study 117380 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117380?search=study&search_terms=117380#rs